CLINICAL TRIAL: NCT00958932
Title: Telecommunication Enhanced Asthma Management
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Bruce Bender, Professor of Pediatrics, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HL084067-01A1 (NIH)
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Speech recognition (TEAM intervention) (Experimental): Parents randomized to the intervention received speech recognition phone calls if their child's medication refill was overdue.
  Interventions: Behavioral: Speech recognition
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Speech recognition — The TEAM intervention is a program to increase communication with families, provide feedback to families about their refill adherence, assess asthma symptoms, deliver health communication messages, encourage parents to ask questions of asthma care managers, and facilitate refilling ICS prescription. Speech recognition calls will be tailored to specific situations including new or re-issued ICS prescriptions, failure to fill an initial prescription, failure to refill, or failure to refill following an ED visit, hospitalization, or oral steroid burst resulting from an asthma exacerbation.
  Other Names: usual care
  Arms: Speech recognition (TEAM intervention)

SUMMARY:
The primary aim of this project is to conduct a randomized practical clinical trial within a large health maintenance organization to test a telephone intervention designed to improve adherence to daily asthma medications and thereby improve asthma outcomes. The investigators hypothesize that adherence with inhaled corticosteroid medications in the TEAM intervention group will be greater than in the usual care group.

DETAILED DESCRIPTION:
Asthma affects more than 15 million people in the United States. Inhaled corticosteroids (ICS), the ranking treatment-of-choice, are safe and highly efficacious in controlled trials, but adherence to ICS medications in real-world settings is poor in all patient groups, especially low-income and minority patients who experience the most morbidity from asthma. Children and adults with asthma take less than half of their prescribed ICS medication. One study found that only 44% of ICS prescriptions for children with asthma were filled. Even the most effective medications have little value if not taken as prescribed. Decreasing use of ICS has been repeatedly linked to poor asthma control and increasing health care utilization.

We will conduct a randomized, practical clinical trial to test the impact of a communication enhancement program for parents of 3-12 year old children with asthma in the largest health maintenance organization (HMO) within Colorado. Research in this setting has the significant advantage of not only establishing the utility of a behavior-changing strategy, but at the same time demonstrating that the strategy can be applied in a large healthcare system and sustained over time. The proposed intervention will be referred to here as the Telecommunication Enhanced Adherence Management (TEAM) program. This proposal builds upon ongoing efforts within Kaiser Permanente of Colorado (KPCO), the participating HMO, to use automated telecommunication technology to prevent diabetes, reduce cardiac risk, reduce calorie consumption, and increase exercise adherence, with the introduction of an intervention to increase adherence with daily ICS therapy. Speech Recognition (SR), the telecommunication technology used in this trial, has not previously been employed to promote adherence in a population of children treated for asthma within a large HMO. TEAM creates a theory-based enhanced communication program using SR with support from asthma care manager nurses. The Asthma Care Manager program already exists within KPCO, but with SR the frequency and quality of communication with parents is expected to improve significantly, resulting in more ICS medication refills, better persistence in ICS use, and improved asthma outcomes. Through SR calls, parents will be reminded and motivated about the importance of continued daily use of ICS medications, asked about their child's recent asthma symptoms, and given the opportunity to receive a call back from an asthma care manager or to place a request for a medication refill.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 year old children with asthma requiring daily corticosteroid

Exclusion Criteria:

* sibling already in study
* physician excludes from participation
* non English Speaking

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1187 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G Bender, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Bender BG, Cvietusa PJ, Goodrich GK, Lowe R, Nuanes HA, Rand C, Shetterly S, Tacinas C, Vollmer WM, Wagner N, Wamboldt FS, Xu S, Magid DJ. Pragmatic trial of health care technologies to improve adherence to pediatric asthma treatment: a randomized clinical trial. JAMA Pediatr. 2015 Apr;169(4):317-23. doi: 10.1001/jamapediatrics.2014.3280. PMID 25664620
- [Derived] Bender BG, Cvietusa PJ, Goodrich GK, King DK, Shoup JA. Adapting adaptive design methods to accelerate adoption of a digital asthma management intervention. Transl Behav Med. 2023 Apr 3;13(3):149-155. doi: 10.1093/tbm/ibac093. PMID 36689336

RESULTS

PARTICIPANT FLOW:
Groups:
- Speech Recognition (TEAM Intervention): Speech recognition: The speech recognition intervention was designed to contact families overdue for a refill and encourage greater ICS adherence, personalizing the conversation with information in the EHR while using language designed to activate parents. Families randomized to the Intervention group received one of three speech recognition call types up to eleven times within each year depending on patterns of overdue refills. All routine clinical services, including telephone availability of asthma nurses and pharmacy staff, were available to both Intervention and Usual Care families.
- Speech Recognition (Usual Care): Speech recognition: Automated, speech recognition telephone calls
Period: Overall Study
Arm/Group | Speech Recognition (TEAM Intervention) | Speech Recognition (Usual Care)
Started | 590 | 597
Completed | 452 | 447
Not Completed | 138 | 150

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Speech Recognition (TEAM Intervention) | Speech Recognition (Usual Care) | Total
Number analyzed (Participants) | 590 | 597 | 1187
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (2.6) | 8.2 (2.2) | 8.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 195 | 424
  Male | 361 | 402 | 763
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 9 | 17
  Asian | 17 | 23 | 40
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 80 | 74 | 154
  White | 330 | 339 | 669
  More than one race | 139 | 146 | 285
  Unknown or Not Reported | 13 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 146 | 146 | 292
  Not Hispanic or Latino | 431 | 449 | 880
  Unknown or Not Reported | 13 | 2 | 15
Region of Enrollment [Number; unit: participants]
  United States | 590 | 597 | 1187

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: The primary outcome of this study, adherence, was expressed as a mean proportion of days covered (PDC) over 24 months. The PDC was calculated as the total number of ICS days supplied divided by the period for which the medication was prescribed. Calculation of the PDC was adjusted to account for the supply that would extend beyond the end of the study period. Comparisons were adjusted for baseline PDC, which was calculated as the ratio of number of days a patient had possession of medication divided by the number of days enrolled 1 year prior to randomization.
Time Frame: 12 months
Population: The 899 participants remaining in the final analysis represent those who remained in the insurance network at 24 months post-randomization.
Measure: Mean (95% Confidence Interval); unit: Proportion of Days Covered
Arm/Group | Speech Recognition (TEAM Intervention) | Speech Recognition (Usual Care)
Number analyzed (Participants) | 452 | 447
Proportion of Days Covered | .445 [.433 to .457] | .355 [.344 to .366]

2. Secondary Outcome: Emergency Care Visits Per Person-Year
Description: Asthma-related emergency care events were compared between the two study groups. In health insurance data, individual records often do not cover the entire period of study because people may leave the insurance network seeking new coverage, or after moving, etc. However, this partial data is still usable when pooled to calculate numbers of events of interest per person-year. For example, one person may only be in the study for six months, and they may log an emergency room. Another person may be in the study for 18 months and log no visits. Put together, the two participants log two person years of data (6 months + 18 months = 24 months = 2 person-years in the study) and between the two of them they log one emergency room visit, which results in an outcome of 0.5 emergency care visits, on average, per person-year of data available. This measure of central tendency is calculated for the two study groups to permit comparison.
Time Frame: Per one year of person-time
Measure: Number (95% Confidence Interval); unit: Number of visits per person-year
Arm/Group | Speech Recognition (TEAM Intervention) | Speech Recognition (Usual Care)
Number analyzed (Participants) | 452 | 447
Number of visits per person-year | 0.06 [.05 to .07] | 0.04 [.03 to .05]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Speech Recognition (TEAM Intervention) | Speech Recognition (Usual Care)
Serious Adverse Events (participants affected / at risk) | 0/590 | 0/597
Other Adverse Events (participants affected / at risk) | 0/590 | 0/597

LIMITATIONS AND CAVEATS:
A potential limitation to this study is that the most poorly adherent patients may have been excluded from the study since eligible patients were required to have made at least 1 Inhaled Corticosteroid fill in the 6 months prior to enrollment. An additional limitation may be non-applicability of the intervention to practices without an Electronic Health Record (EHR) or with an EHR that is different from the one used at Kaiser Permanente Colorado (KPCO).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No